CLINICAL TRIAL: NCT05832060
Title: Comparing the Efficacy of tDCS and tRNS to Improve Reading Skills in Children and Adolescents With Dyslexia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Deny Menghini, Head of Psychology Unit, Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2639_OPBG_2021
Record Dates: First submitted 2023-04-03; First posted 2023-04-27 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Developmental Dyslexia
Keywords: Children; Adolescents; tRNS; transcranial random noise stimulation; tDCS; transcranial direct current stimulation; neurodevelopmental disorders; non-invasive brain stimulation; transcranial electrical stimulation; EEG; reading abilities
MeSH Terms: conditions — Dyslexia; Neurodevelopmental Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- tDCS, tRNS, Sham (Experimental): 1. Active left anodal/right cathodal tDCS over TPC
  2. Active tRNS over bilateral TPC
  3. Sham tRNS or tDCS over bilateral TPC
  Interventions: Device: Active tDCS; Device: Active tRNS; Device: Sham tRNS or tDCS
- tDCS, Sham, tRNS (Experimental): 1. Active left anodal/right cathodal tDCS over TPC
  2. Sham tRNS or tDCS over bilateral TPC
  3. Active tRNS over bilateral TPC
  Interventions: Device: Active tDCS; Device: Active tRNS; Device: Sham tRNS or tDCS
- tRNS, tDCS, Sham (Experimental): 1. Active tRNS over bilateral TPC
  2. Active left anodal/right cathodal tDCS over TPC
  3. Sham tRNS or tDCS over bilateral TPC
  Interventions: Device: Active tDCS; Device: Active tRNS; Device: Sham tRNS or tDCS
- tRNS, Sham, tDCS (Experimental): 1. Active tRNS over bilateral TPC
  2. Sham tRNS or tDCS over bilateral TPC
  3. Active left anodal/right cathodal tDCS over TPC
  Interventions: Device: Active tDCS; Device: Active tRNS; Device: Sham tRNS or tDCS
- Sham, tDCS, tRNS (Experimental): 1. Sham tRNS or tDCS over bilateral TPC
  2. Active left anodal/right cathodal tDCS over TPC
  3. Active tRNS over bilateral TPC
  Interventions: Device: Active tDCS; Device: Active tRNS; Device: Sham tRNS or tDCS
- Sham, tRNS, tDCS (Experimental): 1. Sham tRNS or tDCS over bilateral TPC
  2. Active tRNS over bilateral TPC
  3. Active left anodal/right cathodal tDCS over TPC
  Interventions: Device: Active tDCS; Device: Active tRNS; Device: Sham tRNS or tDCS

INTERVENTIONS:
Device: Active tDCS — Active tDCS will be delivered over TPC for a stimulation session. The anodal electrode will be placed on the left TPC, T7/TP7 position according to the 10-20 International EEG 10-20 System for electrode placement. The cathodal electrode will be placed on the right TPC, T8/TP8 position. Intensity will be set at 1 mA, the duration of stimulation will be 20 min.
Device: Active tRNS — Active tRNS will be delivered to bilateral TPC for a stimulation session. The electrodes will be placed on the left and right TPC, respectively T7/TP7 and T8/TP8 position, at 0.75 mA (100-500 Hz) for 20 min.
Device: Sham tRNS or tDCS — Sham tRNS or tDCS will be delivered over bilateral TPC for a stimulation session. The same electrodes placement as well as the stimulation set-up will be used as in the active stimulation conditions, but the current will be applied for 30 s and will be ramped down without the participants awareness.

SUMMARY:
The present study grounds on the absence of evidence-based treatment in individuals with developmental dyslexia (DD). At this topic, the present study will explore the potential effect of transcranial random noise stimulation (tRNS) and transcranial direct current stimulation (tDCS) over bilateral temporo-parietal cortex (TPC), cerebral areas usually disrupted in individuals with DD.

The investigators hypothesized that active tRNS and tDCS over TPC will boost reading skills in children and adolescents with DD. On the contrary, sham (placebo) tRNS and tDCS over TPC will not have significant effect in improving reading skills. Further, both active and sham tRNS and tDCS will be safe and well tolerated.

DETAILED DESCRIPTION:
The study design is within-subject, randomized stratified, double blind, placebo-controlled.

A group of children and adolescents with DD will be selected and exposed to three different conditions with an interval-session of at least 6 days: 1. tRNS over bilateral TPC; 2. anodal tDCS over left TPC (cathode over right TPC); 3. sham tRNS or tDCS. During stimulation (both real and sham), participants will undergo a concomitant reading task.

In this project, the investigators will work to understand whether a brain-based intervention, with the use of tRNS and tDCS, can improve the outcome of individuals with DD.

The protocol will allow the investigators to:

* comparing the efficacy of tDCS and tRNS over TPC in improving reading abilities,
* comparing the safety and tolerability of tDCS and tRNS in children and adolescents.

The investigator's overarching goal is to provide a scientific foundation for devising new rehabilitation strategies in DD, based on the two most used brain stimulation techniques in pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents with dyslexia (DSM-5, APA 2013)
* IQ ≥ 85

Exclusion Criteria:

* Having a comorbidity with an important medical conditions;
* Having neurological diseases;
* Having Epilepsy o family history of epilepsy;
* Receiving a treatment for dyslexia in the previous three months before the baseline screening.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Text reading accuracy (Experimental reading task) | during procedure
  Change from baseline in text reading accuracy during Active tDCS and Active tRNS sessions than during Sham tDCS and Sham tRNS sessions. Text reading accuracy is considered as the percentage (%) of accuracy and computed as the ratio between the number of correctly read stimuli and the total number of stimuli presented multiplied by 100.

SECONDARY OUTCOMES:
Text reading speed (Experimental reading task) | during procedure
  Change from baseline in text reading speed during Active tDCS and Active tRNS sessions than during Sham tDCS and Sham tRNS sessions. Text reading speed is considered as the syllables/seconds ratio and calculated dividing the total number of syllables pronounced by the total time spent to complete the reading (in seconds).
Experimental reading task: high-frequency word reading accuracy | during procedure
  Change from baseline in high-frequency word reading accuracy during Active tDCS and Active tRNS sessions than during Sham tDCS and Sham tRNS sessions. High-frequency word reading accuracy is considered as the percentage (%) of accuracy and computed as the ratio between the number of correctly read stimuli and the total number of stimuli presented multiplied by 100.
Experimental reading task: high-frequency word reading speed | during procedure
  Change from baseline in high-frequency word reading speed during Active tDCS and Active tRNS sessions than during Sham tDCS and Sham tRNS sessions. High-frequency word reading speed is considered as the syllables/seconds ratio and calculated dividing the total number of syllables pronounced by the total time spent to complete the reading (in seconds).
Experimental reading task: low-frequency word reading accuracy | during procedure
  Change from baseline in low-frequency word reading accuracy during Active tDCS and Active tRNS sessions than during Sham tDCS and Sham tRNS sessions. Low-frequency word reading accuracy is considered as the percentage (%) of accuracy and computed as the ratio between the number of correctly read stimuli and the total number of stimuli presented multiplied by 100.
Experimental reading task: low-frequency word reading speed | during procedure
  Change from baseline in low-frequency word reading speed during Active tDCS and Active tRNS sessions than during Sham tDCS and Sham tRNS sessions. Low-frequency word reading speed is considered as the syllables/seconds ratio and calculated dividing the total number of syllables pronounced by the total time spent to complete the reading (in seconds).
Experimental reading task: non-word reading accuracy | during procedure
  Change from baseline in non-word reading accuracy during Active tDCS and Active tRNS sessions than during Sham tDCS and Sham tRNS sessions. Non-word reading accuracy is considered as the percentage (%) of accuracy and computed as the ratio between the number of correctly read stimuli and the total number of stimuli presented multiplied by 100.
Experimental reading task: non-word reading speed | during procedure
  Change from baseline in non-word reading speed during Active tDCS and Active tRNS sessions than during Sham tDCS and Sham tRNS sessions. Non-word reading speed is considered as the syllables/seconds ratio and calculated dividing the total number of syllables pronounced by the total time spent to complete the reading (in seconds).

CONTACTS AND LOCATIONS:
Locations (1):
- Bambino Gesù Hospital and Research Institute, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shaywitz BA, Shaywitz SE, Pugh KR, Mencl WE, Fulbright RK, Skudlarski P, Constable RT, Marchione KE, Fletcher JM, Lyon GR, Gore JC. Disruption of posterior brain systems for reading in children with developmental dyslexia. Biol Psychiatry. 2002 Jul 15;52(2):101-10. doi: 10.1016/s0006-3223(02)01365-3. PMID 12114001
- [Result] Temple E, Deutsch GK, Poldrack RA, Miller SL, Tallal P, Merzenich MM, Gabrieli JD. Neural deficits in children with dyslexia ameliorated by behavioral remediation: evidence from functional MRI. Proc Natl Acad Sci U S A. 2003 Mar 4;100(5):2860-5. doi: 10.1073/pnas.0030098100. Epub 2003 Feb 25. PMID 12604786
- [Result] Hoeft F, McCandliss BD, Black JM, Gantman A, Zakerani N, Hulme C, Lyytinen H, Whitfield-Gabrieli S, Glover GH, Reiss AL, Gabrieli JD. Neural systems predicting long-term outcome in dyslexia. Proc Natl Acad Sci U S A. 2011 Jan 4;108(1):361-6. doi: 10.1073/pnas.1008950108. Epub 2010 Dec 20. PMID 21173250
- [Result] Hoeft F, Hernandez A, McMillon G, Taylor-Hill H, Martindale JL, Meyler A, Keller TA, Siok WT, Deutsch GK, Just MA, Whitfield-Gabrieli S, Gabrieli JD. Neural basis of dyslexia: a comparison between dyslexic and nondyslexic children equated for reading ability. J Neurosci. 2006 Oct 18;26(42):10700-8. doi: 10.1523/JNEUROSCI.4931-05.2006. PMID 17050709
- [Result] Shaywitz SE, Shaywitz BA, Pugh KR, Fulbright RK, Constable RT, Mencl WE, Shankweiler DP, Liberman AM, Skudlarski P, Fletcher JM, Katz L, Marchione KE, Lacadie C, Gatenby C, Gore JC. Functional disruption in the organization of the brain for reading in dyslexia. Proc Natl Acad Sci U S A. 1998 Mar 3;95(5):2636-41. doi: 10.1073/pnas.95.5.2636. PMID 9482939
- [Result] Bakker DJ. Treatment of developmental dyslexia: a review. Pediatr Rehabil. 2006 Jan-Mar;9(1):3-13. doi: 10.1080/13638490500065392. PMID 16352500
- [Result] Simos PG, Fletcher JM, Bergman E, Breier JI, Foorman BR, Castillo EM, Davis RN, Fitzgerald M, Papanicolaou AC. Dyslexia-specific brain activation profile becomes normal following successful remedial training. Neurology. 2002 Apr 23;58(8):1203-13. doi: 10.1212/wnl.58.8.1203. PMID 11971088
- [Result] Stuss DT. The future of cognitive neurorehabilitation. Neuropsychol Rehabil. 2011 Oct;21(5):755-68. doi: 10.1080/09602011.2011.605590. Epub 2011 Sep 27. PMID 21950776
- [Result] Looi CY, Lim J, Sella F, Lolliot S, Duta M, Avramenko AA, Cohen Kadosh R. Transcranial random noise stimulation and cognitive training to improve learning and cognition of the atypically developing brain: A pilot study. Sci Rep. 2017 Jul 5;7(1):4633. doi: 10.1038/s41598-017-04649-x. PMID 28680099
- [Result] Nitsche MA, Schauenburg A, Lang N, Liebetanz D, Exner C, Paulus W, Tergau F. Facilitation of implicit motor learning by weak transcranial direct current stimulation of the primary motor cortex in the human. J Cogn Neurosci. 2003 May 15;15(4):619-26. doi: 10.1162/089892903321662994. PMID 12803972
- [Result] Fregni F, Boggio PS, Nitsche M, Bermpohl F, Antal A, Feredoes E, Marcolin MA, Rigonatti SP, Silva MT, Paulus W, Pascual-Leone A. Anodal transcranial direct current stimulation of prefrontal cortex enhances working memory. Exp Brain Res. 2005 Sep;166(1):23-30. doi: 10.1007/s00221-005-2334-6. Epub 2005 Jul 6. PMID 15999258
- [Result] Cattaneo Z, Pisoni A, Papagno C. Transcranial direct current stimulation over Broca's region improves phonemic and semantic fluency in healthy individuals. Neuroscience. 2011 Jun 2;183:64-70. doi: 10.1016/j.neuroscience.2011.03.058. Epub 2011 Apr 6. PMID 21477637
- [Result] Schlaug G, Renga V, Nair D. Transcranial direct current stimulation in stroke recovery. Arch Neurol. 2008 Dec;65(12):1571-6. doi: 10.1001/archneur.65.12.1571. PMID 19064743
- [Result] Baker JM, Rorden C, Fridriksson J. Using transcranial direct-current stimulation to treat stroke patients with aphasia. Stroke. 2010 Jun;41(6):1229-36. doi: 10.1161/STROKEAHA.109.576785. Epub 2010 Apr 15. PMID 20395612
- [Result] Monti A, Cogiamanian F, Marceglia S, Ferrucci R, Mameli F, Mrakic-Sposta S, Vergari M, Zago S, Priori A. Improved naming after transcranial direct current stimulation in aphasia. J Neurol Neurosurg Psychiatry. 2008 Apr;79(4):451-3. doi: 10.1136/jnnp.2007.135277. Epub 2007 Dec 20. PMID 18096677
- [Result] Schneider HD, Hopp JP. The use of the Bilingual Aphasia Test for assessment and transcranial direct current stimulation to modulate language acquisition in minimally verbal children with autism. Clin Linguist Phon. 2011 Jun;25(6-7):640-54. doi: 10.3109/02699206.2011.570852. Epub 2011 Jun 1. PMID 21631313
- [Result] Vines BW, Norton AC, Schlaug G. Non-invasive brain stimulation enhances the effects of melodic intonation therapy. Front Psychol. 2011 Sep 26;2:230. doi: 10.3389/fpsyg.2011.00230. eCollection 2011. PMID 21980313
- [Result] Miniussi C, Rossini PM. Transcranial magnetic stimulation in cognitive rehabilitation. Neuropsychol Rehabil. 2011 Oct;21(5):579-601. doi: 10.1080/09602011.2011.562689. Epub 2011 Jun 24. PMID 21462081
- [Result] Ferrucci R, Mameli F, Guidi I, Mrakic-Sposta S, Vergari M, Marceglia S, Cogiamanian F, Barbieri S, Scarpini E, Priori A. Transcranial direct current stimulation improves recognition memory in Alzheimer disease. Neurology. 2008 Aug 12;71(7):493-8. doi: 10.1212/01.wnl.0000317060.43722.a3. Epub 2008 Jun 4. PMID 18525028
- [Result] Rufener KS, Krauel K, Meyer M, Heinze HJ, Zaehle T. Transcranial electrical stimulation improves phoneme processing in developmental dyslexia. Brain Stimul. 2019 Jul-Aug;12(4):930-937. doi: 10.1016/j.brs.2019.02.007. Epub 2019 Feb 13. PMID 30826318
- [Result] Heth I, Lavidor M. Improved reading measures in adults with dyslexia following transcranial direct current stimulation treatment. Neuropsychologia. 2015 Apr;70:107-13. doi: 10.1016/j.neuropsychologia.2015.02.022. Epub 2015 Feb 19. PMID 25701796
- [Result] Costanzo F, Varuzza C, Rossi S, Sdoia S, Varvara P, Oliveri M, Giacomo K, Vicari S, Menghini D. Evidence for reading improvement following tDCS treatment in children and adolescents with Dyslexia. Restor Neurol Neurosci. 2016;34(2):215-26. doi: 10.3233/RNN-150561. PMID 26890096
- [Result] Poreisz C, Boros K, Antal A, Paulus W. Safety aspects of transcranial direct current stimulation concerning healthy subjects and patients. Brain Res Bull. 2007 May 30;72(4-6):208-14. doi: 10.1016/j.brainresbull.2007.01.004. Epub 2007 Jan 24. PMID 17452283
- [Result] Lang N, Siebner HR, Ward NS, Lee L, Nitsche MA, Paulus W, Rothwell JC, Lemon RN, Frackowiak RS. How does transcranial DC stimulation of the primary motor cortex alter regional neuronal activity in the human brain? Eur J Neurosci. 2005 Jul;22(2):495-504. doi: 10.1111/j.1460-9568.2005.04233.x. PMID 16045502
- [Result] Lindenberg R, Renga V, Zhu LL, Nair D, Schlaug G. Bihemispheric brain stimulation facilitates motor recovery in chronic stroke patients. Neurology. 2010 Dec 14;75(24):2176-84. doi: 10.1212/WNL.0b013e318202013a. Epub 2010 Nov 10. PMID 21068427
- [Result] Schlaug G, Marchina S, Norton A. From Singing to Speaking: Why Singing May Lead to Recovery of Expressive Language Function in Patients with Broca's Aphasia. Music Percept. 2008 Apr 1;25(4):315-323. doi: 10.1525/MP.2008.25.4.315. PMID 21197418
- [Result] Rubio-Morell B, Rotenberg A, Hernandez-Exposito S, Pascual-Leone A. [The use of noninvasive brain stimulation in childhood psychiatric disorders: new diagnostic and therapeutic opportunities and challenges]. Rev Neurol. 2011 Aug 16;53(4):209-25. Spanish. PMID 21780073
- [Result] Jancke L, Cheetham M, Baumgartner T. Virtual reality and the role of the prefrontal cortex in adults and children. Front Neurosci. 2009 May 1;3(1):52-9. doi: 10.3389/neuro.01.006.2009. eCollection 2009 May. PMID 19753097
- [Result] Mattai A, Miller R, Weisinger B, Greenstein D, Bakalar J, Tossell J, David C, Wassermann EM, Rapoport J, Gogtay N. Tolerability of transcranial direct current stimulation in childhood-onset schizophrenia. Brain Stimul. 2011 Oct;4(4):275-80. doi: 10.1016/j.brs.2011.01.001. Epub 2011 Feb 1. PMID 22032743
- [Result] Brunoni AR, Amadera J, Berbel B, Volz MS, Rizzerio BG, Fregni F. A systematic review on reporting and assessment of adverse effects associated with transcranial direct current stimulation. Int J Neuropsychopharmacol. 2011 Sep;14(8):1133-45. doi: 10.1017/S1461145710001690. Epub 2011 Feb 15. PMID 21320389
- [Result] Terney D, Chaieb L, Moliadze V, Antal A, Paulus W. Increasing human brain excitability by transcranial high-frequency random noise stimulation. J Neurosci. 2008 Dec 24;28(52):14147-55. doi: 10.1523/JNEUROSCI.4248-08.2008. PMID 19109497
- [Result] Cappelletti M, Gessaroli E, Hithersay R, Mitolo M, Didino D, Kanai R, Cohen Kadosh R, Walsh V. Transfer of cognitive training across magnitude dimensions achieved with concurrent brain stimulation of the parietal lobe. J Neurosci. 2013 Sep 11;33(37):14899-907. doi: 10.1523/JNEUROSCI.1692-13.2013. PMID 24027289
- [Result] Chaieb L, Antal A, Pisoni A, Saiote C, Opitz A, Ambrus GG, Focke N, Paulus W. Safety of 5 kHz tACS. Brain Stimul. 2014 Jan-Feb;7(1):92-6. doi: 10.1016/j.brs.2013.08.004. Epub 2013 Sep 13. PMID 24064065
- [Result] Costanzo F, Menghini D, Caltagirone C, Oliveri M, Vicari S. High frequency rTMS over the left parietal lobule increases non-word reading accuracy. Neuropsychologia. 2012 Sep;50(11):2645-51. doi: 10.1016/j.neuropsychologia.2012.07.017. Epub 2012 Jul 20. PMID 22820638
- [Result] Costanzo F, Rossi S, Varuzza C, Varvara P, Vicari S, Menghini D. Long-lasting improvement following tDCS treatment combined with a training for reading in children and adolescents with dyslexia. Neuropsychologia. 2019 Jul;130:38-43. doi: 10.1016/j.neuropsychologia.2018.03.016. Epub 2018 Mar 14. PMID 29550525
- [Result] Costanzo F, Varuzza C, Rossi S, Sdoia S, Varvara P, Oliveri M, Koch G, Vicari S, Menghini D. Reading changes in children and adolescents with dyslexia after transcranial direct current stimulation. Neuroreport. 2016 Mar 23;27(5):295-300. doi: 10.1097/WNR.0000000000000536. PMID 26848997
- [Result] Fertonani A, Pirulli C, Miniussi C. Random noise stimulation improves neuroplasticity in perceptual learning. J Neurosci. 2011 Oct 26;31(43):15416-23. doi: 10.1523/JNEUROSCI.2002-11.2011. PMID 22031888
- [Result] Snowball A, Tachtsidis I, Popescu T, Thompson J, Delazer M, Zamarian L, Zhu T, Cohen Kadosh R. Long-term enhancement of brain function and cognition using cognitive training and brain stimulation. Curr Biol. 2013 Jun 3;23(11):987-92. doi: 10.1016/j.cub.2013.04.045. Epub 2013 May 16. PMID 23684971
- [Result] Turkeltaub PE, Benson J, Hamilton RH, Datta A, Bikson M, Coslett HB. Left lateralizing transcranial direct current stimulation improves reading efficiency. Brain Stimul. 2012 Jul;5(3):201-207. doi: 10.1016/j.brs.2011.04.002. Epub 2011 May 5. PMID 22305346
- [Result] Linkersdorfer J, Lonnemann J, Lindberg S, Hasselhorn M, Fiebach CJ. Grey matter alterations co-localize with functional abnormalities in developmental dyslexia: an ALE meta-analysis. PLoS One. 2012;7(8):e43122. doi: 10.1371/journal.pone.0043122. Epub 2012 Aug 20. PMID 22916214
- [Result] Gandiga PC, Hummel FC, Cohen LG. Transcranial DC stimulation (tDCS): a tool for double-blind sham-controlled clinical studies in brain stimulation. Clin Neurophysiol. 2006 Apr;117(4):845-50. doi: 10.1016/j.clinph.2005.12.003. Epub 2006 Jan 19. PMID 16427357
- [Result] Ambrus GG, Paulus W, Antal A. Cutaneous perception thresholds of electrical stimulation methods: comparison of tDCS and tRNS. Clin Neurophysiol. 2010 Nov;121(11):1908-14. doi: 10.1016/j.clinph.2010.04.020. Epub 2010 May 14. PMID 20471313
- [Result] Berger I, Dakwar-Kawar O, Grossman ES, Nahum M, Cohen Kadosh R. Scaffolding the attention-deficit/hyperactivity disorder brain using transcranial direct current and random noise stimulation: A randomized controlled trial. Clin Neurophysiol. 2021 Mar;132(3):699-707. doi: 10.1016/j.clinph.2021.01.005. Epub 2021 Jan 27. PMID 33561725
- [Result] Breitling C, Zaehle T, Dannhauer M, Tegelbeckers J, Flechtner HH, Krauel K. Comparison between conventional and HD-tDCS of the right inferior frontal gyrus in children and adolescents with ADHD. Clin Neurophysiol. 2020 May;131(5):1146-1154. doi: 10.1016/j.clinph.2019.12.412. Epub 2020 Jan 24. PMID 32029377
- [Result] Paulesu E, Danelli L, Berlingeri M. Reading the dyslexic brain: multiple dysfunctional routes revealed by a new meta-analysis of PET and fMRI activation studies. Front Hum Neurosci. 2014 Nov 11;8:830. doi: 10.3389/fnhum.2014.00830. eCollection 2014. PMID 25426043
- [Result] Richlan F, Kronbichler M, Wimmer H. Structural abnormalities in the dyslexic brain: a meta-analysis of voxel-based morphometry studies. Hum Brain Mapp. 2013 Nov;34(11):3055-65. doi: 10.1002/hbm.22127. Epub 2012 Jun 19. PMID 22711189
- [Result] Vandermosten M, Boets B, Wouters J, Ghesquiere P. A qualitative and quantitative review of diffusion tensor imaging studies in reading and dyslexia. Neurosci Biobehav Rev. 2012 Jul;36(6):1532-52. doi: 10.1016/j.neubiorev.2012.04.002. Epub 2012 Apr 17. PMID 22516793